CLINICAL TRIAL: NCT07095452
Title: Phase 2/3, Multicenter, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Etentamig and Daratumumab (Etentamig+D) Compared to Daratumumab, Lenalidomide, and Dexamethasone (DRd) in Subjects With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Brief Title: A Study to Assess A Change in Disease Activity and Adverse Events of Intravenous Etentamig and Daratumumab (Etentamig+D) Compared to Daratumumab, Lenalidomide, and Dexamethasone (DRd) in Adult Participants With Newly Diagnosed Multiple Myeloma Not Eligible for Transplant
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: IFM (Intergroupe Français du Myélome); PETHEMA (Program for the Study and Treatment of Haematological Malignances) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-586; 2025-520897-21 (Other: EUCT)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Etentamig; Daratumumab; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 2: Etentamig + Daratumumab Dose A (Experimental): Participants will receive etentamig dose A in combination with daratumumab until the recommended phase 3 dose (RP3D), as part of the approximately 16 year study duration.
  Interventions: Drug: Etentamig; Drug: Daratumumab
- Phase 2: Etentamig + Daratumumab Dose B (Experimental): Participants will receive etentamig dose B in combination with daratumumab until the RP3D, as part of the approximately 16 year study duration.
  Interventions: Drug: Etentamig; Drug: Daratumumab
- Phase 2: Etentamig + Daratumumab Dose C (Experimental): Participants will receive etentamig dose C in combination with daratumumab until the RP3D, as part of the approximately 16 year study duration.
  Interventions: Drug: Etentamig; Drug: Daratumumab
- Phase 3: Etentamig + Daratumumab RP3D (Experimental): Participants will receive etentamig at the RP3D in combination with daratumumab, as part of the approximately 16 year study duration.
  Interventions: Drug: Etentamig; Drug: Daratumumab
- Phase 3: Daratumumab, Lenalidomide, and Dexamethasone (DRd) (Experimental): Participants will receive DRd, as part of the approximately 16 year study duration.
  Interventions: Drug: Lenalidomide; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion
  Arms: Phase 2: Etentamig + Daratumumab Dose A; Phase 2: Etentamig + Daratumumab Dose B; Phase 2: Etentamig + Daratumumab Dose C; Phase 3: Etentamig + Daratumumab RP3D
Drug: Lenalidomide — Oral Capsule
  Arms: Phase 3: Daratumumab, Lenalidomide, and Dexamethasone (DRd)
Drug: Daratumumab — Subcutaneous Injection
Drug: Dexamethasone — Oral Tablet
  Arms: Phase 3: Daratumumab, Lenalidomide, and Dexamethasone (DRd)
Drug: Dexamethasone — IV Injection
  Arms: Phase 3: Daratumumab, Lenalidomide, and Dexamethasone (DRd)

SUMMARY:
Multiple myeloma (MM) is a cancer of the blood's plasma cells. The cancer is typically found in the bones and bone marrow (the spongy tissue inside of the bones) and can cause bone pain, fractures, infections, weaker bones, and kidney failure. This is a study to determine the adverse events, change in disease activity, and pharmacokinetics of Etentamig in adult participants with MM.

Etentamig is an investigational drug being developed for the treatment of MM. This study is broken into 2 phases; phase 2 with 3 study arms and phase 3 with 2 study arms. Participants in phase 2 will receive 1 of 3 doses of etentamig in combination with daratumumab. Participants in phase 3 will receive etentamig at RP3D in combination with daratumumab, or daratumumab, lenalidomide, and dexamethasone (DRd). Around 660 adult participants with MM will be enrolled at approximately 155 sites worldwide

Participants in phase 2 will receive 1 of 3 doses of etentamig as intravenous (IV) infusions, combination with subcutaneous (SC) injections of daratumumab. Participants in phase 3 will receive RP3D doses of etentamig as IV infusions, combination with SC injections of daratumumab, or SC injections of daratumumab, capsules of lenalidomide, and tablet/ IV injections of dexamethasone (DRd). The study duration is approximately 16 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed new diagnosis of multiple myeloma (NDMM) according to the International Myeloma Working Group (IMWG) diagnostic criteria, and per investigator's judgement, participant is not suitable to receive high-dose chemotherapy and stem cell transplantation due to factors likely to have a negative impact on tolerability of high dose chemotherapy and autologous stem cell transplants (ASCT).
* IMWG Myeloma Frailty Index Score of >= 1
* All participants must have measurable disease per central laboratory with at least 1 of the following assessed within 28 days prior to enrollment:

  * Serum M-protein >= 0.5 g/dL (>= 5 g/L).
  * Urine M-protein >= 200 mg/24 hours.
  * Serum free light chain (FLC) >= 100 mg/L (>= 10 mg/dL) (involved light chain) and an abnormal serum kappa lambda ratio only for participants without measurable serum or urine M-protein.

Exclusion Criteria:

* Prior or current systemic therapy or stem cell transplant (SCT) for multiple myeloma or any plasma cell dyscrasia other than short course of corticosteroids
* Participant treated with any investigational treatment within 30 days or 5 half-lives of the treatment (whichever is longer) prior to the first dose of study treatment or is currently enrolled in another clinical study
* Participant who has known active central nervous system involvement of MM.
* Participant who has history of clinically significant renal, neurologic, psychiatric, endocrine, metabolic, immunologic, pulmonary, or hepatic disease within the last 6 months that, in the investigator's opinion, would adversely affect the participant's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2042-01 (Estimated); Study Completion 2042-01 (Estimated)

PRIMARY OUTCOMES:
Phase 2 and 3: Percentage of Participants with Adverse Events (AE)s | Up to Approximately 16 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Phase 2: Change in Clinical Activity | Up to Approximately 52 weeks
  Clinical activity is defined as change in response rates [Overall Response Rate (ORR), Complete Response (CR) or Better, Very Good Partial Response (VGPR), Partial Response (PR)] as determined International Myeloma Working Group (IMWG (2016).
Phase 3: Minimal Residual Disease (MRD) Negative CR Rate | Up to Approximately 52 weeks
  MRDnegCR rate, is defined as the percentage of participants who have achieved stringent complete response (sCR) or CR as assessed by independent review committee (IRC) and have negative MRD defined at 10^-5 threshold as assessed by next generation sequencing (NGS).
Phase 3: Progression-Free Survival (PFS) | Up to Approximately 130 Months
  PFS is defined as the duration from the date of randomization to the date of confirmed disease progression (PD) determined by IRC per IMWG (2016) response criteria, or death, whichever occurs first.

SECONDARY OUTCOMES:
Phase 2: MRD Negative CR Rate | Up to Approximately 52 Weeks
  MRDnegCR rate, is defined as the percentage of participants who have achieved sCR or CR and have negative MRD defined at 10^-5 threshold as assessed by NGS.
Phase 2: PFS | Up to Approximately 130 Months
  PFS is defined as the duration from the date of randomization to the date of confirmed disease progression (PD) determined by IRC per IMWG (2016) response criteria, or death, whichever occurs first.
Phase 2: Sustained MRD Negativity Rate | Up to Approximately 12 Months
  The rate of sustained MRD-negativity is defined as the percentage of participants with maintenance of MRD negativity status in bone marrow confirmed >=12 months apart prior to initiation of new anti-MM therapy.
Phase 2: Area Under the Serum Concentration-Time Curve (AUC) | Up to Approximately 12 Months
  Area under the plasma concentration-time curve (AUC).
Phase 2: Overall Survival (OS) | Up to Approximately 16 Years
  OS is defined as the duration from the date of randomization to the date of the participant's death.
Phase 2: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | Up to Approximately 16 Years
  Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs)
Phase 2: Maximum Observed Serum Concentration (Cmax) | Up to Approximately 12 Months
  Maximum observed serum concentration (Cmax).
Phase 2: Time to Cmax (Time to Maximum Observed Concentration, Tmax) | Up to Approximately 12 Months
  Time to Cmax.
Phase 2: Positive Anti-Drug Antibodies (ADAs) | Up to Approximately 90 days after the last dose of study treatment
  Positive ADAs.
Phase 2: Negative ADAs | Up to Approximately 90 days after the last dose of study treatment
  Negative ADAs.
Phase 2: Neutralizing Anti-Drug Antibodies (NAbs) | Up to Approximately 90 days after the last dose of study treatment
  Neutralizing anti-drug antibodies (NAbs).
Phase 3: OS | Up to Approximately 16 Years
  OS is defined as the duration from the date of randomization to the date of the participant's death.
Phase 3: Sustained MRD Negativity Rate | Up to Approximately 12 Months
  The rate of sustained MRD-negativity is defined as the percentage of participants with maintenance of MRD negativity status in bone marrow confirmed >=12 months apart prior to initiation of new anti-MM therapy.
Phase 3: Rate of >= CR | Up to Approximately 12 Months
  The rate of >= CR is defined as the percentage of participants who achieve a sCR or CR determined by IMWG (2016) response criteria, per IRC assessment, prior to the initiation of new anti-myeloma therapy.
Phase 3: Rate of >= VGPR or Better | Up to Approximately 12 Months
  The rate of >= VGPR is defined as the percentage of participants who achieve a VGPR or better determined by IMWG (2016) response criteria, per IRC assessment, prior to the initiation of new anti-myeloma therapy.
Phase 3: ORR | Up to Approximately 52 Weeks
  ORR is defined as percentage of participants with a response of PR or better per IMWG criteria.
Phase 3: Time to Response (TTR) | Up to Approximately 12 Months
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by IMWG criteria as assessed by investigator.
Phase 3: Duration of Response (DOR) | Up to Approximately 16 Years
  DOR is defined as the number of days from the day the response criteria are met to the date that disease progression.
Phase 3: Time-to-Progression (TTP) | Up to Approximately 16 Years
  Time to progression is defined as the number of days from the date of study drug start to the date of the first documented disease progression or relapse.
Phase 3: Event Free Survival (EFS) | Up to Approximately 16 Years
  EFS will be measured as the number of days between the initiation of the studied line of therapy and disease progression, or refractory disease, or death.
Phase 3: Progression-Free Survival on Subsequent Therapy (PFS2) | Up to Approximately 16 Years
  PFS2 is defined as the duration from the date of randomization to the date of confirmed disease progression or death on the next line of therapy.
Phase 3: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | Up to Approximately 16 Years
  Incidence, severity, seriousness, and causality of TEAEs
Phase 3: Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Physical Functioning Score | Up to Approximately 16 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Subjects rate items on a 4- point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Phase 3: Change from Baseline in EORTC QLQ-C30 Global Health Status/QoL Score | Up to Approximately 16 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Subjects rate items on a 4- point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Phase 3: Change from Baseline and Time to Deterioration in the Remaining Scales and Items of EORTC QLQ-C30 | Up to Approximately 16 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Subjects rate items on a 4- point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Phase 3: Symptomatic AEs as Assessed by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to Approximately 16 Years
  PRO-CTCAE includes 124 items representing 78 symptomatic toxicities drawn from the CTCAE. PRO-CTCAE items evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. All questions employ a 7-day recall period and are scored from 0 to 4 (or 0/1 for absent/present).
Phase 3: Overall Bother Due to Treatment Side Effects as Assessed by the Functional Assessment of Cancer Therapy-General (FACT-G) GP5 | Up to Approximately 16 Years
  The FACT-G GP5 Item is a part of the FACT-G which is a 27-item questionnaire that measures four domains of health-related quality of life (HRQOL) in cancer patients: physical, social, emotional and functional well-being. The FACT-G GP5 item ("I am bothered by side effects of treatment") is used to assess overall treatment tolerability in patients by assessing the overall side effect impact on patients. This item is rated on a 5-point Likert scale from "not at all" to "very much.".
Phase 3: Change from Baseline in Patient Global Impression of Severity (PGIS) Scores | Up to Approximately 16 Years
  The PGIS scale asks the patient to assess their overall QoL, as well as difficulty of doing physical activities due to MM over the past 7 days. Each item employs a 5-point Likert scale from "not at all" to "very much."
Phase 3: Change from Baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) Scores | Up to Approximately 16 Years
  The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (7):
  - Colorado Blood Cancer Institute /ID# 279080, Denver, Colorado
  - Fort Wayne Medical Oncology And Hematology /ID# 278141, Fort Wayne, Indiana
  - Willamette Valley Cancer Institute and Research Center /ID# 278721, Eugene, Oregon
  - SCRI Oncology Partners /ID# 278353, Nashville, Tennessee
  - Texas Oncology - The Woodlands /ID# 278726, The Woodlands, Texas
  - Texas Oncology - Northeast Texas /ID# 278725, Tyler, Texas
  - Blue Ridge Cancer Care - Roanoke /ID# 278722, Roanoke, Virginia
- Japan (3):
  - Matsuyama Red Cross Hospital /ID# 278660, Matsuyama, Ehime
  - Tokai University Hospital /ID# 278157, Isehara, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 278156, Kyoto, Kyoto

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-586